CLINICAL TRIAL: NCT04949802
Title: A Prospective Single Center Clinical Study for Femtosecond Laser Glaucoma Surgery Using the ViaLase Laser
Brief Title: Glaucoma Surgery Using the ViaLase Laser System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vialase, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIA-001
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Glaucoma; Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Masking Description: observer-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Laser (Experimental): Treated with ViaLase Laser
  Interventions: Device: ViaLase Laser

INTERVENTIONS:
Device: ViaLase Laser — ViaLase Laser System to create an aperture through the trabecular meshwork for the reduction of IOP in subjects with primary open-angle glaucoma

SUMMARY:
Prospective, single-center, multi-cohort clinical trial of ViaLase Laser for the reduction of IOP in patients with open angle glaucoma.

DETAILED DESCRIPTION:
The purpose of study is to obtain initial evidence of safety of femtosecond laser glaucoma surgery using the ViaLase Laser for the treatment of open angle glaucoma. The ViaLase Laser System is intended to create apertures through the trabecular meshwork to reduce intraocular pressure in patients with open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary open-angle glaucoma (including pigmentary and pseudoexfoliative glaucoma).
2. Glaucomatous visual field defects consistent with optic nerve defects and defined as one or more of the following:

   1. A cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level on the pattern deviation (PD) plot; or
   2. Glaucoma hemi-field test "outside normal limits" Note: Visual field reliability indices (i.e., fixation losses, false positives, and false negatives) should all be less than 33%. For subjects with a screening visual acuity of 20/100 or worse, a visual field is not required, and the above criteria do not need to be met.
3. Nerve abnormality characteristic of glaucoma as evaluated by clinical ophthalmoscopy defined as one or more of the following:

   1. Diffuse thinning, focal narrowing or notching of the optic disc rim especially at inferior or superior poles.
   2. Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at inferior or superior poles.
   3. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue.
4. Subject eye is phakic

   a. If phakic, then the crystalline lens will not have visually significant cataract that is expected to require cataract surgery within next one year. Cataract will be evaluated by using the AREDS clinical lens grading system (ARLNS). Specifically, crystalline lens must have ARLNS grade of ≤ 1.5 for signs of nuclear opalescence, cortical or posterior subcapsular opacities. Lenticular opacities not characterized by the ARLNS grading system shall also be evaluated (e.g. anterior subcapsular cataracts).
5. Mean IOP with medication at screening between 21 mmHg and 35 mmHg, inclusive.
6. Iridocorneal angle anatomy defined as follows:

   1. Trabecular meshwork visible on gonioscopy defined by Shaffer grade ≥ 3.
   2. Normal anatomy as determined by gonioscopy.
7. Light perception or better in the study eye at screening. Note: The non-study eye must not have a Snellen corrected visual acuity (CVA) of worse than 20/200 at screening.
8. Age 45 years or older
9. Available, willing, with sufficient cognitive awareness to comply with examination procedures and schedules.
10. Signed written informed consent.

Exclusion Criteria:

1. Previous glaucoma surgeries including stent implantation or other laser surgeries on study eye.
2. Prior intraocular surgery.
3. Glaucoma types as follows:

   1. Traumatic, uveitic, neovascular, or angle-closure.
   2. Glaucoma associated with vascular disorders.
4. Corneal status as follows:

   1. Any condition that would preclude safe participation in the study or reliable IOP assessments including active inflammation, edema, keratitis, keratoconjunctivitis, keratouveitis.
   2. Clinically significant dystrophy such as bullous keratopathy or Fuch's dystrophy.
   3. Guttata that would preclude safe participation in the study or reliable study assessments.
   4. Anticipated surgery of any type (including LASIK, LASEK, PRK, cataract, etc.) during the study that may alter IOP measurement.
   5. Corneal opacities or disorders that would inhibit visualization of the angle (such as severe arcus senilis).
   6. Central corneal thickness less than 440 microns or greater than 620 microns.
5. Choroid status as follows:

   1. Choroidal detachment
   2. Effusion
   3. Choroiditis
   4. Neovascularization
   5. Any active choroidopathy.
6. Retinal or optic nerve disorders, either degenerative or evolutive, that are not associated with the existing glaucoma condition including: proliferative diabetic retinopathy, central retinal artery occlusion, central retinal vein occlusion, wet age-related macular degeneration, dry age-related macular degeneration (e. g., presence of numerous large drusen associated with disturbance to or elevation of the retinal pigment epithelium), significant retinal pigment epithelial changes or optic atrophy, pathological myopia, red disease.

   Note: Minor diabetic retinopathy or hypertensive retinopathy are permitted.
7. Elevated episcleral venous pressure associated with:

   1. Active thyroid orbitopathy.
   2. Cavernous sinus fistula.
   3. Sturge-Weber syndrome.
   4. Orbital tumors.
   5. Orbital congestive disease.
8. Other ocular conditions as follows:

   1. Sequelae from trauma that would preclude safe participation in the study or reliable study assessments (e.g., chemical burns, blunt trauma, etc.)
   2. Chronic ocular inflammatory disease or presence of active ocular inflammation or infection (e.g., uveitis, iritis, iridocyclitis, retinitis)
   3. Any pathology for which, in the investigator's judgement, the following would be either at risk or contraindicated:

   i. Compliance to elements of the study protocol (e.g., ophthalmic examinations, follow- up visits)

   ii. Subjects with inadequate space in the anterior chamber and/or angle as determined by slit lamp examination and gonioscopy.
9. Subject status as follows:

   1. Uncontrolled systemic disease (e.g. diabetes, hypertension) that could compromise their participation in the study.
   2. Use of systemic medications (either current, within 30 calendar days of screening exam, or anticipated) that may cause an increase in IOP, (e.g. systemic steroids including oral or IV formulation, topical steroids applied on the periorbital surface within ¼" of the external lid margins and oral inhaled steroids). Nasal inhaled steroids are allowed.
   3. Active concurrent enrollment in any investigational trial or previous participation in any investigational trial within 30 days of the screening exam.
   4. Women who are nursing, are pregnant or are of childbearing potential who refuse to use reliable contraception.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Sarayba, MD, Study Director — Vialase, Inc.
Locations (1):
- Semmeweis University Ophthalmology Clinic, Budapest, Hungary

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Laser: Treated with ViaLase Laser
  ViaLase Laser System to create an aperture through the trabecular meshwork for the reduction of IOP in subjects with primary open-angle glaucoma
Period: Overall Study
Arm/Group | Laser
Started | 15; 22 eyes
Completed | 12; 18 eyes
Not Completed | 3; 4 eyes
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | Laser
Number analyzed (Participants) | 15
Number analyzed (eyes) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 15
IOP [Mean (Standard Deviation); unit: mmHg] | 21.3 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP
Description: continuous, mean IOP
Time Frame: 12 months
Population: PP
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Laser
Number analyzed (Participants) | 12
Number analyzed (eyes) | 18
mmHg | 12.7 (2.3)

2. Primary Outcome: Percent Change From Baseline in Intraocular Pressure
Description: Mean Percent Change From Baseline in Intraocular Pressure
Time Frame: 12 months
Population: PP
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Units Other Than Participants: eyes
Arm/Group | Laser
Number analyzed (Participants) | 12
Number analyzed (eyes) | 18
percentage change from baseline | -38.5 (9.8)

3. Secondary Outcome: Number of Eyes That Achieved >=20% IOP Reduction
Description: binary, number of eyes that had an IOP reduction of at least 20% from baseline
Time Frame: 12 months
Population: PP
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Laser
Number analyzed (Participants) | 12
Number analyzed (eyes) | 18
eyes | 18

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Laser
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser (N=15)
COVID 19 (Infections and infestations) | 3 (3) — Hospitalization due to COVID 19, not related to study device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser (N=15)
Cystoid Macular Edema (Eye disorders) | 1 (1) — not related to study device
Anterior Ischemic Optic Neuropathy (Eye disorders) | 1 (1) — not related to study device
BCVA loss >= 2 lines (Eye disorders) | 2 (2) — not related to study device
Visual Field progression, MD loss >=2.5dB (Eye disorders) | 1 (1) — not related to study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04949802/Prot_SAP_000.pdf